CLINICAL TRIAL: NCT00275730
Title: Effects of Indomethacin on Retinal and Choroidal Blood Flow in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 9-11-2004
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Ocular Physiology; Regional Blood Flow
Keywords: indometacine; retinal blood flow; choroidal blood flow
MeSH Terms: interventions — Indomethacin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: indometacine (drug) effect on ocular blood flow

SUMMARY:
Prostaglandins (PG) are known to alter regional ocular blood flow and exhibit vasoactive properties in isolated ocular blood vessels. A variety of animal experiments indicate that endogenous PGs play a role in the regulation of retinal (RBF) and choroidal (ChBF) blood flow. There is also evidence that the prostaglandin pathway is involved in the activation of NO production in humans, however, the mechanisms for interactions between PG and NO in ocular vasculature are still unclear.

Animal studies suggest that retinal and choroidal blood flow decrease after administration of indomethacin (a nonspecific cyclooxygenase inhibitor). More recently, it has been shown that indomethacin injected intravenously decreased optic nerve oxygen tension and reduced the CO2 reactivity. This is probably the result of decreased blood flow through vasoconstriction of vessels in the optic nerve. Systemic administration of indomethacin also diminishes cerebral, renal and mesenteric blood flow by an unknown mechanism. However, no clinical trials exist so far investigating the effects of indomethacin on ocular blood flow. Therefore, the aim of this study is to investigate the effect of indomethacin on ocular blood flow in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropy less than 3 dpt

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Retinal and choroidal blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria